CLINICAL TRIAL: NCT01832194
Title: Use of Botox to Treat Scrotal Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAN_BTX
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2013-04

CONDITIONS: Scrotal Pain
Keywords: Scrotal pain; Botox
MeSH Terms: interventions — Botulinum Toxins, Type A; onabotulinum toxin A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Botox (Experimental): Botox:
  A concentrated dose of Onabotulinum Toxin A of 100 units dissolved in 2 cc of 2% xylocaine for a one-time injection.
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox
  Other Names: Onabotulinum Toxin A

SUMMARY:
There are no previous reports on the use of Onabotulinum Toxin A to treat men with scrotal pain that we found published. We propose a pilot study to use Botox to block the testicular nerves on a group of 15 men with chronic scrotal pain who have failed the standard medical therapy. The men must have had temporary relief from a testicular cord block using marcaine. Before and 1 month, 3 months and 6 months after the Onabotulinum Toxin A injection, the men would be asked to fill in visual analog scales for pain, a quality of life assessment, a depression index (MDI) and Chronic Epididymitis Symptom Index (CESI). They will also be subject to sensory testing of the scrotum before, after 1 month, 3 moths and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Have nociceptive scrotal pain,
* Have no identifiable, reversible causes for the scrotal pain
* Have failed standard medical therapy
* Have responded temporarily to cord blocks

Exclusion Criteria:

* Are interested in trying to conceive with their partners in the next 6 months,
* Have any local infection near the site of the injections,
* Have had an allergic reaction to Botox in the past,
* Are unable to provide informed consent
* Have a history of motor neuron disease or neurogenic bladder
* Who have hemostatic disorder or who are taking aspirin, Coumadin (warfarin), Xarelto (rivaroxaban) or other blood thinners

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in pain | 6 months after entering in trial
  Change in pain is measured by visual analog scales for pain, a quality of life assessment, a depression index (MDI) and Chronic Epididymitis Symptom Index (CESI) before therapy and 1, 3 and 6 months post therapy. In addition, physical examination of the testis and epididymis and sensory testing of the skin of the scrotum and anterior thigh before the therapy and 1, 3 and 6 months post therapy. The sensory testing will be the patients' subjective reporting of the sensation felt with light touch (normal, decreased, increased or painful) and pin prick (decreased, normal or increased) in the skin of the scrotum and anterior thigh of the treated side (the side where the therapy was used) compared to the untreated side (where no therapy was used).

CONTACTS AND LOCATIONS:
Overall Officials: Keith Jarvi, MD, Principal Investigator — Mount Sinai Hospital, Canada
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada